CLINICAL TRIAL: NCT03535753
Title: Safety and Efficacy Evaluation of Decitabine With R-GDP on Refractory or Relapsed NHL Patients
Brief Title: Safety and Efficacy Evaluation of Decitabine With R-GDP
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Immunochina Medical Science & Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M201791
Record Dates: First submitted 2018-05-14; First posted 2018-05-24 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2017-09

CONDITIONS: NHL
MeSH Terms: interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Decitabine and R-GDP (Experimental): ALL patients will be treated with Decitabine and R-GDP
  Interventions: Drug: Decitabine and R-GDP

INTERVENTIONS:
Drug: Decitabine and R-GDP — Decitabine and R-GDP
  Other Names: DR

SUMMARY:
Assessment of the Safety and efficacy of Administering decitabin plus R-GDP to NHL patients

DETAILED DESCRIPTION:
RR NHL patients will be treated with decitabin plus R-GDP , safety and efficacy will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed or refractory Non-Hodgkin's lymphoma(NHL) patiens.
2. Eastern Cooperative Oncology Group(ECOG) score 0-2
3. Expected survival >3 months
4. Measurable disease.

Exclusion Criteria:

1. Patients who needs treatment with immunosuppressive agents
2. Hematosepsis or Uncontrolled active infection
3. History of epilepsy or other CNS disease.
4. Active hepatitis B , hepatitis C or HIV infection or any other uncontrolled active infection.
5. Pregnancy or breast-feeding women.
6. Any uncontrolled medical disorders that the researchers considered are not suitable to participate the clinical trial.
7. Any situation that would increase dangerousness of subjects or disturb the outcome of the clinical study according to the researcher's evaluatio

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
OS | 2 years
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Hongmei Jing, MD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking university third hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No